CLINICAL TRIAL: NCT04676711
Title: A First-in-human, Randomized, Double-blinded, Placebo- Controlled, Two-part Study to Assess Safety/Tolerability and Pharmacokinetics of Single- and Multiple-ascending Doses and Food Effect of GFH312 in Healthy Subjects
Brief Title: A Study of GFH312 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GenFleet Therapeutics (Australia) Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GFH312X3101
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Toxicity; Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Study drug: GFH312 and placebo In part Ia, subjects will be randomized and dosed in different cohorts in single dose. In part Ib, one of the cohorts will selected as food effect cohort with washout period of part Ia.
  In part II, subjects will be randomized and dosed in different cohorts in multiple doses.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GFH312 (Experimental)
  Interventions: Drug: GFH312
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFH312 — Subjects are planned to be dosed in oral tablet, with single and multiple ascending doses
  Arms: GFH312
Drug: Placebo — Subjects are planned to be dosed in oral tablet, with single and multiple ascending doses
  Arms: Placebo

SUMMARY:
GFH312 is a small molecule inhibitor of receptor-interacting serine/threonine protein-1(RIP1) kinase, a key regulator of the TNF-α downstream. RIPK1 can regulate the NF- κB signaling and necroptosis, a type of cell death which can trigger immune response and enhance inflammation. As such, GFH312 represents a novel, selective mechanism for the treatment of inflammatory conditions.

This study is the first administration of GFH312 to humans. The purpose of the study is to evaluate the safety/tolerability and pharmacokinetics in healthy subjects. The intention of this study is to provide confidence in the safety of the molecule to inform progression to further proof-of-concept studies. The dose range proposed in this study is based on a low starting dose escalating to supra-therapeutic doses.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent must be obtained before any assessment is performed.
2. Healthy male and female subjects age 18 to 55 years of age included.
3. Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18-32 kg/m2 inclusive.
4. At screening, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the subject has rested for at least three minutes, and again (when required) after three minutes in the standing position. Sitting vital signs should be within the normal ranges.
5. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant must use highly effective methods of contraception during intercourse while taking drug and for 30 days after stopping study medication; and sexually active males must use a condom, during intercourse while taking drug and for 30 days after stopping study medication.
6. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria

Healthy subjects fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
2. Hemoglobin levels below the lower limit of normal (LLN) as set by the laboratory.
3. An elevated C-reactive protein (CRP) outside of the normal reference range and has clinical significance, or above 10 mg/L.
4. A positive anti-nuclear antibody (ANA) above 1:160 titer.
5. A positive Tuberculosis test.
6. A history of clinically significant ECG abnormalities, or any abnormalities defined in protocol.
7. History of immunodeficiency diseases, including a positive test for HIV antibody.
8. Chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV).
9. Infections requiring parenteral antibiotics within the 6 months prior to Screening.
10. History of any venous thromboembolism, TIA, intracranial hemorrhage, neoplasm, arteriovenous malformation, vasculitis, bleeding disorder, coagulation disorders or screening blood tests that indicate altered coagulability (platelet count, APTT, PT, etc.).
11. History of significant cardiovascular, respiratory, renal, neurological disease.
12. Significant illness which has not resolved within two (2) weeks prior to initial dosing.
13. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
14. Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
15. Known family history or known presence of long QT syndrome, or concomitant use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of study.
16. History of hypersensitivity to any of the study treatments or excipients (e.g., lactose monohydrate) or to drugs of similar chemical classes; and history of anaphylaxis or other significant allergy in the opinion of the Investigator.
17. Donation or loss of 400 ml or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulation.
18. Plasma donation (>400 mL) within 14 days prior to first dosing.
19. Use of any prescription drugs, herbal supplements (including Silybum marianum and Valeriana officinalis), within two weeks prior to initial dosing, and/or over-the- counter (OTC) medication, dietary supplements (vitamins included) within one weeks prior to initial dosing.
20. Smokers of more than two per week. Urine cotinine levels will be measured during screening, and urine cotinine ≥ 500 ng/ml will exclude a subject.
21. History of drug abuse or unhealthy alcohol use within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during screening.
22. History of recreational cannabis use within four weeks prior to dosing, or evidence of such use as indicated by the laboratory assays conducted during screening.
23. Participant is unwilling to refrain from strenuous exercise (including weightlifting) from 7 days prior to admission to the site until completion of the final Follow-up visit.
24. With a plan to receive vaccination with a live vaccine within 4 weeks prior to the first dosing or within 4 weeks of the last dosing; With a plan to receive COVID-19 vaccination within 2 weeks prior to the first dosing or within 1 week of the last dosing.
25. Exposure to any significantly immune suppressing drug (including experimental therapies as part of a clinical trial) within the 4 months prior to screening or 5 half-lives, whichever is longer.
26. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, or twice the duration of the biological effect of the investigational product, whichever is longer; or longer if required by local regulations.
27. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
28. (Part Ⅱ only) Score 'yes' on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or 'yes' on any item of the Suicidal Behavior section, except for the 'Non-Suicidal Self-Injurious Behavior' (item also included in the Suicidal Behavior section), if this behavior occurred in the past 2 years. Or history of drug abuse or mental disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Safety /Tolerability of GFH312 (adverse events) | approximately 45 days
  Incidence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No